CLINICAL TRIAL: NCT05349019
Title: A Natural History Study of Patients With Parkinson's Disease (PD) Caused by the p.Gly2019Ser (G2019S) Pathogenic Mutation of the Leucine-Rich Repeat Kinase 2 (LRRK2) Gene
Brief Title: A Natural History Study of Patients With G2019S LRRK2 Parkinson's Disease
Status: Terminated | Type: Observational
Why Stopped: Sponsor stopped the study
Sponsor: Escape Bio, Inc. (Industry)
Collaborators: Momentum Pharma (Industry); Science 37 (Industry)
Responsible Party: Sponsor
Other Study IDs: ESBG2019S-001
Record Dates: First submitted 2022-04-14; First posted 2022-04-27 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-08

CONDITIONS: Patients With Parkinson's Disease (PD) Caused by the p.Gly2019Ser (G2019S) Pathogenic Mutation of the Leucine-Rich Repeat Kinase 2 (LRRK2) Gene
Keywords: G2019S LRRK2 mutation
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Part A/Sub Cohort A1: 15 healthy participants 18-35 years of age
  Interventions: Other: Observational
- Part A/Sub Cohort A2: 15 healthy participants 65-80 years of age
  Interventions: Other: Observational
- Part A/Sub Cohort A3: Control group age and sex matched to the PD participants in Part B of the study
  Interventions: Other: Observational
- Part B: 60 participants with a confirmed diagnosis of Parkinson's disease and a heterozygous G2019S mutation in the LRRK2 gene
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is an observational study to investigate the natural history of G2019S LRRK2 PD using traditional and digital methodology (digital phenotyping). Study conduct will be decentralized (at home as much as possible) consisting of two parts: Part A with Healthy Volunteers (HV) participants and Part B in patients with G2019S LRRK2 PD.

SUMMARY:
To characterize using a participant centered decentralized (at home) study featuring wearable technology and telemedicine to study disease change over time in patients with PD caused by the G2019S mutation in the LRRK2 gene and to identify a clinical endpoint(s) for disease modifying experimental therapy trials.

ELIGIBILITY:
Part A Inclusion Criteria (Healthy Volunteers)

Individuals eligible to participate in Part A of this study will meet all the following criteria:

1. Willing and able to provide informed consent after the nature of the study has been explained
2. 18-35 years of age inclusive at Screening (sub cohort A1) or 65-80 years of age inclusive at Screening (sub cohort A2)
3. Willing and able to comply with all study procedures
4. Sub cohort A3 participants must match the age ± 0.5 years and sex of match participant in Part B
5. Participant must be healthy as per the investigator's assessment with no underlying clinically significant diseases (participants with hypertension, diabetes, hypercholesterolemia, and other chronic diseases associated with aging but not thought to interfere with the performance of the mTUG or other study measures may be allowed after consultation with the Medical Monitor)
6. Participant must be able to use the Technology as described in the protocol
7. Have access to a minimum indoor space of 6 meters by 2 meters (or approximately 20 feet by 7 feet) to carry out the mTUG
8. Agree to retain the same level of activity throughout the study and not have plans to stop/start or increase or decrease any exercise programs
9. Have reliable access to working WiFi internet or willingness to use a provided cellular internet connection device
10. Agree to refrain from all alcohol and cannabinoid products within 24 hours prior to performing the mTUG assessment (i.e., three non consecutive days during study Week two, and Weeks two and three of the run in period)

Part A Exclusion Criteria (Healthy Volunteers)

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

1. History of mobility, gait, or ambulation problems (defined as mobility limitations that impact walking on a daily basis)
2. History of neurological disease
3. Any elective surgery planned during the study duration, approximately 12-15 months from Screening
4. History of significant head injury within the past 5 years (head injury with loss of consciousness or requiring greater than 24 hours in hospital in relation to head injury)
5. History of alcohol use disorder or other substance abuse disorder (excluding tobacco use), according to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) in the past 10 years
6. Body Mass Index (BMI) (calculated from self reported height and weight) of greater than 35
7. Pregnant or planning to become pregnant in the next 24 months
8. Has a concurrent disease or condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety

Part B Inclusion Criteria (PD Patients)

Individuals eligible to participate in Part B of this study must meet all the following criteria:

1. Willing and able to provide informed consent after the nature of the study has been explained
2. Willing and able to comply with all study procedures
3. Have confirmed diagnosis of PD documented in medical records according to UK Brain Bank criteria
4. Confirmed G2019S mutation(s) in the LRRK2 gene either by evidence recorded in medical record with report from accredited laboratory, or through another accredited genetic testing program, or other partner laboratory. Up to 10 participants with homozygous mutations may be enrolled in addition to the 60 participants with heterozygous mutation
5. Hoehn and Yahr Scale Score 1-3
6. Physically and cognitively able to complete protocol specified tasks independently or with some assistance
7. If assistance is required for completion of tasks (e.g., help with the Technology), a caregiver or volunteer must be fully available to assist the participant for the duration of the study
8. Ability to complete the mTUG without the use of a cane or walker and without a personal assistant
9. Ability to complete the mTUG which is not impacted by comorbidities (e.g., participant should not have underlying, clinically significant cardiac or respiratory disease, or musculoskeletal disease). Non-progressive diseases of these organ systems must be approved by the Medical Monitor prior to enrollment; for example, mild to moderate osteoarthritis may be allowable
10. Have access to a minimum indoor space of 6 meters by 2 meters (or approximately 20 feet by 7 feet) to carry out the mTUG
11. A helper or participant is required to be present during the performance of mTUG, if the participant has had more than one fall in the past 12 months
12. The participant's general health status is acceptable for participation in the study (per their physician)
13. Working WiFi internet or willing to use a provided cellular internet connection device
14. Participant must agree to refrain from all alcohol and cannabinoid products within 24 hours prior to performing the mTUG (i.e., three non consecutive days during study Week two, and Weeks two and four of the run in period)

Part B Exclusion Criteria (PD Patients)

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

1. Any mobility, gait, or ambulation problems other than those related to PD
2. Any deep brain stimulation in situ or planned during the study duration, approximately 12-15 months from Screening
3. Any planned changes in physiotherapy or exercise therapy
4. Planned initiation of, or changes in, cognitive behavioral therapy
5. Any elective planned surgery during the study duration, approximately 12-15 months from Screening
6. History of significant head injury within the past 5 years (head injury with loss of consciousness or requiring greater than 24 hours in hospital in relation to head injury)
7. History of frequent falls (classified as one fall every 1 month)
8. Any other genetic PD causing mutations, for example, a pathogenic GBA mutation
9. History of alcohol use disorder or other substance abuse disorder (excluding tobacco use), according to the DSM-5 in the past 10 years
10. Any other serious concomitant diseases unrelated to PD (e.g., other neurological diseases of any kind, renal failure, liver failure, active cancer)
11. BMI (calculated from self reported height and weight) of greater than 35
12. Pregnant or planning to become pregnant in the next 24 months
13. Has a concurrent disease or condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Part A (Healthy Volunteers): Healthy participants aged 18-80 years of age
  * Part B (Patients with Parkinson Disease): Participants with PD caused by the G2019S pathogenic mutation of the LRRK2 gene
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Compare the change over 12 months in the modified Timed Up and Go (mTUG) test | 12 months
  To compare the change over 12 months in the modified Timed Up and Go (mTUG) test, or subitems of the mTUG, recorded by video and a smartphone sensor application between participants with PD caused by the G2019S pathogenic mutation of the LRRK2 gene, and age and sex matched healthy control cohort

SECONDARY OUTCOMES:
Evaluate the change over 12 months in linear velocity parameter in ambulation and gait. | 12 months
  To evaluate the change over 12 months in parameter ambulation and gait including linear velocity measured in meters/second.
Evaluate the change over 12 months in stride length parameter in ambulation and gait. | 12 months
  To evaluate the change over 12 months in parameter ambulation and gait including stride length measured in meter.
Evaluate the change over 12 months in cadence parameter in ambulation and gait. | 12 months
  To evaluate the change over 12 months in parameter ambulation and gait including cadence measured in steps per minute.
Evaluate the change over 12 months in double support parameter in ambulation and gait. | 12 months
  To evaluate the change over 12 months in parameter ambulation and gait including double support time as measured in milliseconds in a real world setting using a digital insole device.

CONTACTS AND LOCATIONS:
Overall Officials: Carrolee Barlow, MD, PhD, Study Chair — Escape Bio, Inc.
Locations (1):
- Science 37, Culver City, California, United States

REFERENCES:
- [Background] Bright JM, Carlisle HJ, Toda AMA, Murphy M, Molitor TP, Wren P, Andruska KM, Liu E, Barlow C. Differential Inhibition of LRRK2 in Parkinson's Disease Patient Blood by a G2019S Selective LRRK2 Inhibitor. Mov Disord. 2021 Jun;36(6):1362-1371. doi: 10.1002/mds.28490. Epub 2021 Feb 11. PMID 33836114